CLINICAL TRIAL: NCT04589364
Title: A 50-Week Prospective, Double-Blinded, Randomized, Cross-over Design in Multicenter Study of100 Unit of Abobotulinum Toxin Type A (Dysport®) Versus 33.33 Unit of Neubotulinum Toxin Type A (Neuronox®) Injection for Hemifacial Spasm in Thai Patients
Brief Title: Study of Abobotulinum Toxin Versus Neubotulinum Toxin Injection For Hemifacial Spasm in Thai Patients
Acronym: DNHFS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY NO. A-01-2020
Record Dates: First submitted 2020-10-04; First posted 2020-10-19 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Hemifacial Spasm
MeSH Terms: conditions — Hemifacial Spasm

STUDY DESIGN:
Intervention Model Description: A 50-Week Prospective, Double-Blinded, Randomized, Cross-over design in Multicenter Study of 100 unit of Abobotulinum Toxin Type A (Dysport) versus 33.33 unit of Neubotulinum Toxin Type A (Neuronox) Injection For Hemifacial Spasm in Thai Patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- abobotulinum toxin A (Experimental): Abobotulinum Toxin Type A (Dysport) dose was investigated:
  dose: 100 units ( various units each site depend on clinical )
  Interventions: Drug: Injection botulinum toxin A ( Dysport 100 unit or Neuronox 33.33 unit)
- neubotulinum toxin A (Experimental): Neubotulinum Toxin Type A (Neuronox) dose was investigated:
  dose: 33.33 units ( various units each site depend on clinical )
  Interventions: Drug: Injection botulinum toxin A ( Dysport 100 unit or Neuronox 33.33 unit)

INTERVENTIONS:
Drug: Injection botulinum toxin A ( Dysport 100 unit or Neuronox 33.33 unit) — injection of toxin on facial muscle

SUMMARY:
A 50-Week Prospective, Double-Blinded, Randomized, Cross-over design in Multicenter Study of 100 unit of Abobotulinum Toxin Type A (Dysport®) versus 33.33 unit of Neubotulinum Toxin Type A (Neuronox®) Injection for Hemifacial Spasm in Thai Patients, designed gor comparing the effectiveness of Total intensity score after 4. 12. 16 and 24 weeks of treatment and to compare the long-term safety of the injections. Abobotulinum toxin A (Dysport *) dose 100 units compared ot neubotulinum toxin A injection (Neuronox / Neuronox®) dose 33.33 units. that it si non-inferiority (non-inferiority) ni the treatment of hemifacial spasm after administration of the drug ni the 0, 12" ,26", and 38" weeks ni the treatment of patients with hemi facial spasm, with a wash out period of 2 weeks between treatments. By proving the non-inferiority of Total intensity score at ,4 ,8 and12 week after treatment which calculated by severity score and duration of facial muscle spasm (hour per day)., as well as severity score and duration of functional impairment (hour per day) recorded for 4,8, and 21 weeks after each treatment between 33.33 unit of Neubotulinum Toxin Type A(Neuronox*) and 100 unit of Abobotulinum Toxin Type A (Dysport*)

DETAILED DESCRIPTION:
There were two treatment arms in crossover designed study and the interest was on the comparison of total intensity score, duration of hemifcial spasm and duration of functional impairment in each pre- and post- treatment outcomes of (Dysport®) and (Neuronox®) , two pair-wised comparisons pre and post treatment after ,4- 8- and 12-week scale were carried out. For each of the pair-wise comparison, 2-sided p-value was used ot ensure that the overall Type I error-0.05. Beta error 80% (Multiple repeated analysis and general linear model may be analyses) in the efficacy of treatment. Two-sided exact p-values were reported in the efficacy analyses. Demographic and safety analyses were based on the summary of descriptive statistics.This study had a washout period of 2 weeks because there was a study on hemifacial spasm that Botulinum toxin A loses its effect before 12 weeks from a study of its action by Katalin Bihari and colleagues who found that Onabotulinumtoxin A (Botox®) has a duration of action in hemifacial spasm of 64.3 days compared to Abobotulinum toxin A (Dysport ®) has a duration of action ni hemifacial spasm of 41.8 days 5 (reference Bihari K. Safety, effectiveness, and duration of effect of Botox after switching from disport for blepharospasm, cervical dystonia and hemifacial spasm. Curr Med Res Opin 2005 Mar; 21(3):433-8). Another 5 studies as follows: Lolekha (2017) found that Onabotulinumtoxin A (Botox®) had a duration of action ni hemifacial spasm of 72.24 days. A, Yoshimura (1992) found that Onabotulinumtoxin A (Botox ®) has a duration of action in hemifacial spasm of 84 days. A, Rieder (2007) found that Onabotulinumtoxin A (Botox®) has a duration of action in hemifacial spasm of 71 days. A, Quagliato (2010) found that Onabotulinumtoxin A(Botox®) There is a duration of action in hemifacial spasm of 89.6 days. A and Kongsaengdao (2012) found that Neu-botulinumtoxin A (Neuronox®) / Abobotulinum Toxin A (Dysport®) had a clear measurement of the duration of action with a Patient diary that recorded symptoms for everyday. The duration of action in hemifacial spasm is 84 days, which has been shown to be no different from Neubotulinum toxin This study required a washout period in this study of 14 days, which si 98 days from the second injection ni V2, which si longer than the longest duration in the double blind randomized controll study. By Quagliato's (2010) which the effect ni hemifacial spasm lasting for 89.6 days.

Studies which not double blinded, randomized studies with a prospective trial design and clearly measured duration of action (Duration of effect from review or estimation or inference) cannot be used as a reference for this study due ot study bias.

Screening Period (-1 to 0 week):

At the screening visit and prior to performance of any study procedures, the investigators would explain the details of the study and the subject would have to sign on the written informed consent, exclusion criteria, and inclusion criteria.

Each subject who was willing to enrol into the study was asked about their medical history as well as their recent and current medications being taken.

Al enrolled subjects were asked to undertake an initial physical examination and had to satisty the criteria for the inclusion /exclusion before being enrolled into the study.

Al patients were asked to complete physical examination, HFS 30, AIMS, SF36, PHQ-9 and CES-D.

Laboratory blood (livers tests, haematology,) examinations, urine pregnancy test) were performed for safety reasons.

Double-Blind Treatment Period Inclusion visit: week -1-0 (V0-1)

After the screening period, al eligible subjects were entered into the treatment period and received either intramuscular injection of 33.33 unit of Neubotulinum Toxin Type A (0.3 ml) or 10 unit of Abobotulinum Toxin Type A. (0.3 ml) The injection was only performed after the subject was confirmed to be eligible against al the inclusion and exclusion criteria. The inclusion visit included the followings examination and tests before injection:

* physical and neurological examinations,
* vital signs,
* weight, urine pregnancy test (if suspected pregnancy or loss regular menstration), CBC, NIR laboratory test ni case of history of abnormal bleeding, HFS 30, AIMS, SF36, PHQ-9 and CES-D, Dispense Patient diary. Concomitant-treatment.

Folow up Visits V2, V3, V4, V5, V6 Visit 2 (V2) Al subject were asked ot complete physical examination, HFS 30, AIMS, SF36, PHQ-9 and CES-D and Patient diary wil be collected and dispense the new Patient diary before injection.

During of the visit, the investigator would conduct before injection:

* physical examination and neurological examination,
* monitoring of the vital signs,
* weight measurements,
* urine pregnancy test (if suspected pregnancy or loss regular menstration),
* Clinical global impression scale (CGIC-physician and patient),
* adverse events,
* Concomitant-treatment. after that, patient will receive either intramuscular injection of 100 unit of Abobotulinum Toxin Type A. (0.3 ml) or 33.33 unit of Neubotulinum Toxin Type A (0.3 ml) as same as Inclusion visit.

Visit 3 (V3) (performed after washout period 2 weeks ) Al subject were asked to complete physical examination, HFS 30, AIMS, SF36, PHQ-9, CGIC and CES-D and Patient diary wil be colected and dispense hte new Patient diary before injection.

During of the visit, the investigator would conduct before injection:

* physical examination and neurological examination,
* monitoring of the vital signs,
* weight measurements,
* urine pregnancy test (if suspected pregnancy or loss regular menstration),
* Clinical global impression scale (CGIC- physician and patient),
* adverse events,
* Concomitant-treatment. after that, patient will receive either intramuscular injection of 50 unit of Neubotulinum Toxin Type A (0.3 ml) or 250 unit of Abobotulinum Toxin Type A. (0.3 ml) by crossover trement with Inclusion visit and visit 2.

Visit 4(V4) All subject were asked to complete physical examination, HFS 30, AIMS, SF36, PHQ-9 and CES-D and Patient diary wil be collected and dispense the new Patient diary.

During of hte visit, the investigator would conduct before injection:

* physical examination and neurological examination,
* monitoring of the vital signs,
* weight measurements,
* urine pregnancy test (if suspected pregnancy or loss regular menstration),
* Clinical global impression scale (CGIC- physician and patient),
* adverse events, after that, patient will receive either intramuscular injection of 33.33 unit of Neubotulinum Toxin Type A(0.3 ml) or 10 unit of Abobotulinum Toxin Type A. (0.3 ml) as same as visit 3.

end Visit (V5) Al subject were asked to complete physical examination, HFS 30, AIMS, SF36, CGIC PHQ-9 and CES-D and Patient diary wil be collected

During of the visit, the investigator would conduct:

* physical examination and neurological examination,
* monitoring of the vital signs,
* weight measurements,
* urine pregnancy test (if suspected pregnancy or loss regular menstration),
* Clinical global impression scale (CGI - physician and patient),
* adverse events,
* Concomitant-treatment. after that patient may received either intramuscular injection of 100 unit of Abobotulinum Toxin Type A. (0.3 ml) or 33.33 unit of Neubotulinum Toxin Type A (0.3 ml) by re-emburstment from national policy.

NOTE: After 4 weeks of treatment of botulinum toxin A injection (weeks 4,16,24,30,42) there was a telephone call, interview, questionnaire HFS 30, AIMS, SF 36, CESD, PHQ9.

Safety folow up Visit (SFV, V6) Al subject were asked ot complete physical examination, by standard botulinum toxin clinic assessment.

During of the visit, the investigator would conduct:

* physical examination and neurological examination,
* monitoring of the vital signs,
* weight measurements,
* urine pregnancy test (if suspected pregnancy or loss regular menstration),, -Clinical global impression scale (CGIC- investigators and patient), adverse events,
* Concomitant-treatment, after that patient may received either 100 unit of Abobotulinum Toxin Type A. (0.3 ml) or 33.33 unit of Neubotulinum Toxin Type A (33.3 ml) by re- emburstment from national policy.

Study Population The study population consisted of male or female subjects, ages ranged between 18-80 years old, diagnosed with hemifacial spasm. These subjects were randomized ot receive 10 unit of Abobotulinum Toxin Type A(Dysport®) and 33.33 unit of Neubotulinum Toxin Type A(Neuronox®) injection in cross-over designed.

Study Duration The study duration was conducted over 62 weeks (-1 to 0 week for the screening period and four of 12-week interval for the double-blind cross over treatment period ( washout period 2 weeks between V2 and V3),and 12 week follow up period.

ELIGIBILITY:
The subjects need to satisfy the following criteria before being allowed to participate ni the study:

1. Volunteers with hemifacial spasm aged 18 to 80 years who may or may not have received Botulinum toxin before.
2. Subjects were diagnosed with hemifacial spasm by a neurologist.
3. Healthy female volunteers of reproductive age must obtain informed consent from the study physician to avoid pregnancy throughout the study by using condoms or an appropriate method of birth control. too Female volunteers will be required to consent ot a urine pregnancy test before entering the study and throughout the study. There will be a pregnancy test using a urine test strip every time fi menstruation is over.
4. Volunteers must be evaluated for reliability ni participating ni the research project and volunteers or relatives can record treatment results. and side effects or drugs used in treatment They are willing to participate in the research project and understand the benefits of participating in the study.
5. The patient has had other normal physical examinations and si able ot undergo a neurological examination as wel as Able ot participate ni physical examinations ot assess symptoms of hemifacial spasm and can cooperate ni completing the AIMS questionnaire, HFS30, 36-item quality of life questionnaire, PHQ9, and the CES-D depression questionnaire.

Exclusion Criteria Criteria for exclusion from the study Patients cannot participate in the research project fi they have the following conditions:

1. The volunteer is pregnant or breastfeeding, or the volunteer si a woman at risk of pregnancy who has not received adequate pregnancy protection.
2. Volunteers who have contraindications or precautions for injection. Botulinum toxin Aor hte need ot use drugs that may cause adverse reactions from Interactions between required drugs and investigational drugs such as aminoglycoside, spectinomycin, polymyxin tetracycline, and lincomycin antibiotics and tubocurarines muscle relaxant.
3. The volunteer has an allergic reaction to hte drug or any substance related to the drug used for treatment.
4. The volunteer is unable or unwilling to participate and follow al details in the research project. or not cooperating in completing questionnaires in the research project.
5. The subject has received any other unregistered drugs or other experimental drugs within the past 6 months. Al types of botulinum toxin are allowed (patients can receive previous treatment with any type of botulinum toxin for more than 14 weeks or 98 The day before the Ist appointment).
6. Volunteers who have been previously selected for this research project.
7. Subjects with a history of botulism or co-morbidities such as neuromuscular junction disease such as myasthenia gravis. or Eaton Lumber Syndrome.
8. Volunteers with other physical diseases or other neurological diseases or psychiatric disorders that may affect treatment. For example, having a history of blood clotting disorders (INR greater than 1.2), low blood platelets. Rheumatoid joint pain, heart attack, coronary artery disease Dementia Any type of psychosis or any other condition or risk factor for adverse reactions that may affect the results of the research.
9. The volunteer has a history of being addicted to or using drugs or narcotics or has a history of allergic reaction to botulinum toxin.
10. Subjects who received planned and treated surgery. throughout the research study period or patients receiving aminoglycosides or culale cannot participate in the research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Total Intensity score | 12 weeks
  Primary efficacy variable Comparesion of pre- and post- treatment at each injection (4 week) and over all after 12- and 24-week scale with 33.33 unit of Neubotulinum Toxin Type A(Neuronox®) and 100 unit of Abobotulinum Toxin Type A(Dysport®); as followings:
  1) Patient diary, the 24 hour HFS diary record for 12 weeks after treatment. Total intensity score at 4, 8, and 12 weeks after treatment [which calculated by severity score and duration of facial muscle spasm (hour per day), as wel as severity score and duration of functional impairment (hour per day) recorded at 4, 8, and 12 weeks after each treatment will be assessed].
Duration of functional impairment per day | 12 weeks
  Primary efficacy variable Comparesion of pre- and post- treatment at each injection (4 week) and over all after 12- and 24-week scale with 33.33 unit of Neubotulinum Toxin Type A(Neuronox®) and 100 unit of Abobotulinum Toxin Type A(Dysport®); as followings:
  1) Patient diary, the 24 hour HFS diary record for 12 weeks after treatment. Duration of functional impairment at 4, 8, and 12 weeks after treatment [which calculated by duration of facial muscle spasm which effect to functional impairment (hour per day),impairment recorded at 4, 8, and 12 weeks after each treatment will be assessed].
Duration of facial muscle spasm per day | 12 weeks
  Primary efficacy variable Comparesion of pre- and post- treatment at each injection (4 week) and over all after 12- and 24-week scale with 33.33 unit of Neubotulinum Toxin Type A(Neuronox®) and 100 unit of Abobotulinum Toxin Type A(Dysport®); as followings:
  1) Patient diary, the 24 hour HFS diary record for 12 weeks after treatment. Duration of facial muscle spasm at 4, 8, and 12 weeks after treatment [which calculated by duration of facial muscle spasm which may or may not effect to functional impairment (hour per day),impairment recorded at 4, 8, and 12 weeks after each treatment will be assessed].

SECONDARY OUTCOMES:
Hemifacial Spasm- 30 Questionnaire | 12 weeks
  Seven subscales (30 items). Mobility 5( items), activity of daily living (5 items) and communication 3( items) are classified sa physical health domain. Emotional wel-being 7( items), stigma 4( items), social support 3( items) and cognition (3 items) are classified as mental health domain at 4, 8, and 12 weeks after each treatment will be assessed].
Abnormal involuntary movement scale | 12 weeks
  Rating sacle of the severity of movements in 7regions, each on a 5points scale and aseparate rating of the overall severity of the abnormal movements, judged on the amplitude of movements, incapacitation postures and positions, including sitting ni chair, opening the mouth, tapping the thumb against each finger, holding the hand out stretched and standing and walking, are included. Dental status is also rated, as the presence or absence of problems with teeth or dentures at 4, 8, and 12 weeks after each treatment will be assessed].
36-item questionnaire scale of general health quality of life | 12 weeks
  eight domains: Physical functioning (PF), Role limitations due to physical health (RP), Role limitations due to emotional problems (RE), Vitality (VT), Mental health (MH), Social functioning (SF), Bodily pain (BP), and General health (GH) at 4, 8, and 12 weeks after each treatment will be assessed].
Center of Epidemiologic study -Depression scale (CES-D) | 12 weeks
  20 item depressive screening scale ( range 0-80 higher score represent worse) at 4, 8, and 12 weeks after each treatment will be assessed].
Patient health Questionnaire - 9 item (PHQ-9) | 12 weeks
  9 item depressive screening scale range between 0-27 higher score represent worse at 4, 8, and 12 weeks after each treatment will be assessed].
The investigator's global assessment of change | 12 weeks
  5 scale evaluate clinical status range from -3 to 3 higher score represent good outcomes at 4, 8, and 12 weeks after each treatment will be assessed].
The patient's global assessment of change | 12 weeks
  5 scale evaluate clinical status range from -3 to 3 higher score represent good outcomes at 4, 8, and 12 weeks after each treatment will be assessed].

CONTACTS AND LOCATIONS:
Locations (4):
- Thailand (4):
  - Rajavithi Hospital, Bangkok
  - Lampang Hospital, Lampang
  - Surat Thani hospital, Surat Thani
  - Sappasitthiprasong Hospital, Ubon Ratchathani

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kongsengdao S, Kritalukkul S. Quality of life in hemifacial spasm patient after treatment with botulinum toxin A; a 24-week, double-blind, randomized, cross-over comparison of Dysport and Neuronox study. J Med Assoc Thai. 2012 Mar;95 Suppl 3:S48-54. PMID 22619887